CLINICAL TRIAL: NCT05252013
Title: The Impact of Broad Bean Hull on Blood Glucose Control and Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 4667
Record Dates: First submitted 2021-12-07; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Healthy; Overweight
Keywords: gut bioavailability; plasma metabolites; faecal metabolites; broad bean hull; high fibre; Vicia faba
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Randomised controlled crossover non-blinded design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plain Bread (Placebo Comparator): Participants will be attending the Human Nutrition Unit in the morning (day 1), following an overnight fast. Fasted blood samples will be taken and one portion of plain bread (122g) served with 25g of jam will be consumed by the volunteers. The meal will be consumed within 15 minutes and postprandial blood samples will be collected. Participants will be provided with the meals for the rest of the day to take away and for days 2 and 3. In total, they will consume 6 plain bread rolls on days 1, 2 and 3 (2 bread rolls/day).
  Interventions: Other: Experimental: Plain Bread
- Broad bean hull bread (Experimental): Participants will be attending the Human Nutrition Unit in the morning, following an overnight fast. Fasted blood samples will be taken and one portion of the bean hull bread (155g) served with 25g of jam will be consumed by the volunteers. The meal will be consumed within 15 minutes and postprandial blood samples will be collected. Participants will be provided with the meals for the rest of the day to take away and for days 2 and 3. In total, they will consume 6 bean hull bread rolls on days 1, 2 and 3 (2 bread rolls/day).
  Interventions: Other: Experimental: Bean Hull Bread

INTERVENTIONS:
Other: Experimental: Bean Hull Bread — The bean hull bread will deliver 21.96 g of fibre. Volunteers will consume a roll of bean hull bread (155g/portion) served with 25g of raspberry jam.
  Other Names: Broad Bean Hull Bread
  Arms: Broad bean hull bread
Other: Experimental: Plain Bread — The control bread will deliver 4.53 g of fibre. Volunteers will consume a roll of plain bread (122g/portion) served with 25g of raspberry jam.
  Other Names: Control Bread
  Arms: Plain Bread

SUMMARY:
This study aims to assess the effects of broad bean hull (BBH) consumption on blood glucose and gut health. Broad bean (Vicia faba) is widely cultivated in Scotland, with the UK being the most significant European producer. The seed coat (hull or testa) is removed during broad bean processing. This is a significant secondary product that is largely discarded. Preliminary work showed that this material is comparable to wheat bran and is rich in fibre (49%) and protein (18%). Additionally, it showed a rich phytochemical profile and lower fat and carbohydrate content than wheat bran. Experiments also showed that BBH inhibited the activity of alpha-amylase and alpha-glucosidase enzymes, suggesting anti-diabetic properties. Overall, these results showed that BBH is a secondary crop product having potential as a functional food for humans. Therefore, the objective of this study is to assess in vivo in humans the physiological and functional effects of BBH. Using an acute phase randomised controlled crossover design, the study will assess how consuming BBH fortified breads affects plasma glucose and gut health. The study will recruit 18 volunteers, normal-overweight, aged 18-75 years, who habitually consume low amounts of fruits and vegetables (≤3 portions/day). The volunteers will attend two identical stand-alone intervention sessions lasting three days each following the screening. The order of the intervention sessions will be randomised. On the day before each intervention session, the participants will provide a baseline faecal sample and have a continuous glucose monitoring sensor (CGMS) attached. They will be also be given a standardised dinner. On the next morning, following a 10-12 hr fast, an indwelling antecubital cannula will be inserted, and a blood sample will be taken for measuring baseline levels of metabolites. The volunteers will be given a standardised portion of the BBH or control bread to consume, and further blood samples taken for the subsequent four hours. Breath samples will also be taken at the same time points for measuring gastric emptying. The volunteers will be provided with all the meals for the rest of the day and the subsequent two days. These will include two portions per day of either the BBH or control bread. The meals will be standardised for energy and macronutrients. The volunteers will be instructed to return to the Human Nutrition Unit on the fourth morning and provide a second faecal sample and remove the CGMS. Blood samples will be analysed for systemic bioavailability and metabolism of test meal components, glucose regulatory hormones and breath samples for quantifying gastric emptying. The faecal samples will be analysed for gut bioavailability and metabolism of test meal components, microbial counts, composition, and water content.

DETAILED DESCRIPTION:
The study aims to confirm in vivo the effects of consuming broad bean hull on blood glucose control and gut health. Although in vitro evidence is promising, its benefits remain confirmed in vivo in humans. No studies have previously attempted to assess the impact of broad bean hull consumption on glycaemic and gut health outcomes in humans. Therefore, this study will be novel and provide useful information on the potential of using BBH as a functional food for human health.

From a health perspective, it is essential to establish the bioavailability and metabolism of dietary constituents in humans. Certain metabolites are absorbed early in the gastrointestinal tract, whereas others are transported to the colon, where they are extensively metabolised by the gut microbiota. This study will characterise the bioactive metabolites present in the plasma and faecal samples obtained. This will inform on their availability to the systemic circulation and their excretion profiles.

Using targeted quantitative analysis (LC-MS and GC-MS), metabolites and their in vivo concentrations will be measured. The principal metabolites analysed will be those produced by the phenylpropanoid pathway and protein and carbohydrate metabolism products. These will include derivatives and metabolites of the simple phenols, benzoic acids, phenolic acids, phenylacetic acids, phenypropionic acids, phenylpyruvic acids, phenyllactic acids, mandellic acids, phenolic dimers, acetophenones, benzaldehydes, cinnamaldehydes, benzyl alcohols, cinnamyl alcohols, indoles, isoflavones, coumarins, chalcones, flavanones, flavones, flavonols, anthocyanidins.

Furthermore, short-chain fatty acids will be analysed in the participants' faecal samples. It has been shown that many of these compounds are bioactive and exhibit anti-oxidant and anti-inflammatory activity at in vivo concentrations. Therefore, these studies will provide important information on bioavailability and metabolism and correlate the indices with health biomarkers.

In addition, compounds such as the carcinogenic heterocyclic amines, genotoxic nitrosamines, indoles, polyamines, bile acids, and other protein metabolites considered detrimental to human health will also be measured. It is likely, the carbohydrate and phytochemical content of plant proteins may also protect against the formation of these toxic and potentially carcinogenic protein by-products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Aged 18-75 years old.
* BMI 23-35 kg/m2
* HbA1c <6.5%
* Total cholesterol ≤ 7 mmol/l

Exclusion Criteria:

* Glucose 6 Phosphate Dehydrogenase deficiency
* Diagnosed for chronic diseases; thyroid disorders, metabolic/genetic diseases, diabetes and disorders of glycaemic control; cardiovascular disease; irritable and inflammatory bowel disorders.
* Women with polycystic ovaries syndrome (PCOS)
* Women who are lactating or breastfeeding, pregnant
* On prescription medications known to affect metabolism, including hormonal contraceptives and thyroid medications, and hormonal replacement therapy
* Have taken a course of antibiotics in the past four weeks
* Allergic/intolerant to foods provided in the study
* Diagnosed for high blood pressure and on prescription medications such as Ramipril
* Alcohol and/or other substance abuse
* Smoking and the use of e-cigarettes, nicotine patches and nicotine gums
* Physically active at a competitive level
* Usually not consuming significantly more than five portions of fruits and vegetables per day
* Poor venous access

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Plasma key bioactive metabolites following the control and bean hull bread consumption | over 4 hours
  The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected postprandial over 4 hours.
  For both the control and test diet, plasma markers of the principal metabolites produced by the phenylpropanoid pathway and products of protein and carbohydrate metabolism will be measured over 4-hour interval and compared with baseline.
Plasma key bioactive metabolites following the control and bean hull bread consumption | Day 4
  The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected on the day. The participants will be provided with plain/bean hull bread rolls to be consumed on day 1 (intervention day), days 2 and 3. Fasted blood samples will be measured on day 4.
  The principal metabolites produced by the phenylpropanoid pathway and products of protein and carbohydrate metabolism following the 3 days consumption of the test and control diet will be measured in fasted plasma of day 4. These metabolites will be compared with the baseline (day 1) and between diets (day 4 vs day 4).
Faecal key bioactive metabolites excretion | Day 4 (post intervention)
  The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, consumed within 15 minutes. Participants will also consume the plain/bean hull bread for days 1, 2, 3. A second faecal sample will be collected on day 4 to assess participants' gut bioavailability of key nutrients and bioactive following the chronic consumption of the plain/bean hull bread rolls.
  The principal metabolites produced by the phenylpropanoid pathway and products of protein and carbohydrate metabolism following the 3 days consumption of the test and control diet will be measured in faecal samples of day 4. These metabolites will be compared with the baseline (day 1) and between diets (day 4 vs day 4).
Determine the effects of consumption bean hull fortified bread on Ghrelin levels | over 4 hours
  To investigate the effect of bean hull bread on ghrelin. The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected on the day. Ghrelin levels will be measured over 4 hours following the consumption of the plain/bean hull bread rolls.
Determine the effects of consumption bean hull fortified bread on GLP-1 levels | over 4 hours
  To investigate the effect of bean hull bread on the hormone GLP-1. The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected on the day. GLP-1 levels will be measured over 4 hours following the consumption of the plain/bean hull bread rolls.
Determine the effects of consumption bean hull fortified bread on glucagon | over 4 hours
  To investigate the effect of bean hull bread on the hormone glucagon. The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected on the day. Glucagon levels will be over 4 hours following the consumption of the plain/bean hull bread rolls.
Determine the effects of consumption bean hull fortified bread on PYY | over 4 hours
  To investigate the effect of bean hull bread on the hormone PYY. The intervention visit will involve a test meal to be consumed by subjects attending the Human Nutrition Unit (HNU) in the morning, following an overnight fast. They will be provided with a meal, which will be consumed within 15 minutes and blood samples will be collected on the day. PYY levels will be measured over 4 hours following the consumption of the plain/bean hull bread rolls.

SECONDARY OUTCOMES:
Postprandial blood glucose responses (recording iAUC and AUC) | Every 5 minutes for 4 hours using a continuous glucose monitor device
  Measuring postprandial glucose levels following the test meals
Postprandial insulin responses (recording iAUC and AUC) | 4 hours and Day 4
  Measuring postprandial insulin levels following the test meals
Microbiota composition change | Day 1 and 4
  Changes in the composition of the microbiota will be based on next-generation sequence analysis of 16S rRNA (ribosomal ribonucleic acid) genes extracted from faecal samples provided by all volunteers
Gastric emptying | 4 hours
  Measuring gastric emptying rate following the consumption of the two test meals

CONTACTS AND LOCATIONS:
Overall Officials: Madalina Neacsu, Principal Investigator — m.neacsu@abdn.ac.uk
Locations (1):
- University of Aberdeen, Rowett Institute, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No